CLINICAL TRIAL: NCT07041866
Title: Impact of the Consumption of Fortified Biscuits on the Iron Status of School-aged Children in a Rural Setting in Kaolack, Central Senegal
Brief Title: Impact of the Consumption of Fortified Biscuits on the Iron Status of School-aged Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universite du Sine Saloum Elhadj Ibrahima Niasse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: USSEIN2024
Record Dates: First submitted 2025-06-19; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: This Study Aimed to Evaluate the Impact of Fortified Biscuit Consumption on the Iron Status of School-aged Children in Rural Kaolack
Keywords: Fortified biscuit, school-aged children, iron status, anemia, nutritional status, Senegal.
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of two parallel groups: an intervention group receiving iron-fortified biscuits and a control group receiving placebo biscuits with similar appearance but without iron-rich ingredients. The intervention lasted for 3 months, and outcomes were assessed before and after the intervention period.
Who Masked: Participant, Outcomes Assessor
Masking Description: In this study, both participants and data collectors were blinded to the group assignments. Participants were unaware whether they were receiving the iron-fortified biscuit or the placebo biscuit, as both were similar in appearance and taste. Additionally, data collectors responsible for anthropometric and biological measurements were not informed of the participants' allocation to ensure objectivity in data collection. However, the study coordinators and investigators were aware of the intervention allocation due to the nature of the study design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): This group included 286 school-aged children (6-16 years) enrolled in a French public elementary school in Keur Socé.
  Interventions: Dietary Supplement: Fortified Biscuit with Local Iron-Rich Ingredients
- Control group (Placebo Comparator): This group consisted of 210 children (aged 6-16 years) from a Franco-Arabic elementary school in the same locality.
  Interventions: Dietary Supplement: Non-Fortified Biscuit

INTERVENTIONS:
Dietary Supplement: Fortified Biscuit with Local Iron-Rich Ingredients — Participants consumed one fortified biscuit per day, five days a week (school days), for a period of three months. The biscuit was formulated using wheat flour, millet, maize, peanut paste, sugar, and was filled with a blend of Moringa oleifera, Hibiscus sabdariffa, Adansonia digitata, and Detarium senegalense-all selected for their high iron and vitamin C content. The iron content was approximately 4 mg per 100 g.
  Arms: Experimental group
Dietary Supplement: Non-Fortified Biscuit — Participants received a placebo biscuit daily for the same period and frequency as the intervention group. The placebo biscuit was visually and texturally identical to the fortified biscuit but did not contain the micronutrient-rich filling.
  Arms: Control group

SUMMARY:
This study aimed to evaluate the impact of fortified biscuit consumption on the iron status of school-aged children in rural Kaolack.

The main question it aims to answer is:

• Does the consumption of iron-fortified biscuits improve the iron status of school-aged children? Researchers compared the iron-fortified biscuit to a placebo (a biscuit similar in appearance but without iron-rich ingredients) to measure its effectiveness.

Participants:

* Consumed either the fortified biscuit or the placebo daily for 3 months
* Took part in data collection after 3 months of biscuit consumption

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 to 16 years
* Enrolled in one of the two selected elementary schools (French or Franco-Arab)
* Availability to participate throughout the 3-month intervention period
* Obtained written informed consent from parent or guardian Verbal assent obtained from the child

Exclusion Criteria:

* Children diagnosed with sickle cell disease (SCD)
* Children currently under iron supplementation or treatment at the start of the study
* Refusal to participate or withdrawal of consent at any time

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 570 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Change in serum ferritin concentration (ng/mL) | At baseline and at 3 months (endline)
Prevalence of iron deficiency | At baseline and at 3 months (endline)

SECONDARY OUTCOMES:
Change in hemoglobin concentration (g/dL) | At baseline and at 3 months (endline)
Prevalence of anemia (mild, moderate, severe) | At baseline and at 3 months (endline
Change in BMI-for-age Z-score (BMIZ-WHO) | At baseline and at 3 months (endline
prevalence of thinness (BMIZ < -2 SD) | At baseline and at 3 months (endline)
C-reactive protein (CRP) concentration | At baseline and at 3 months (endline)
Alpha-1-acid glycoprotein (AGP) concentration | At baseline and at 3 months (endline)

OTHER OUTCOMES:
Sex (male/female) | at baseline
Age of participants | At baseline and at 3 months (endline)

CONTACTS AND LOCATIONS:
Locations (1):
- École Élémentaire de Keur Socé City: Kaolack Country: Senegal, Kaolack, Senegal

IPD SHARING:
Plan to Share IPD: Undecided